CLINICAL TRIAL: NCT02866877
Title: Effects of Augmented Renal Clearance on Pharmacokinetic and Pharmacodynamic Properties of Levetiracetam in Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-1823
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Subarachnoid Hemorrhage
Keywords: augmented renal clearance
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subarachnoid Hemorrhage
  Interventions: Other: Pharmacokinetic modeling

INTERVENTIONS:
Other: Pharmacokinetic modeling — Timed blood draws and urine collections to model drug clearance

SUMMARY:
This study evaluates the pharmacokinetic profile of levetiracetam in critically ill patients who have suffered a subarachnoid hemorrhage. The patients will be evaluated for development of augmented renal clearance and the effects and duration of effects this may have on levetiracetam clearance.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with non-traumatic subarachnoid hemorrhage requiring levetiracetam for seizure prophylaxis or treatment
* Presentation to University of Colorado Hospital within 48 hours of subarachnoid hemorrhage
* Adults ages 18 to 89 years
* Anticipated length of stay ≥ 48 hours
* Informed consent provided by the patient or patient's designated medical proxy

Exclusion Criteria:

* Pregnancy
* Patients receiving renal replacement therapy
* Brain death or imminent brain death expected ≤48 hours
* Patient with history of nephrectomy or renal transplant

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have suffered a non-traumatic subarachnoid hemorrhage requiring strict intake and output monitoring and admission to the neuro-intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Change in systemic levetiracetam clearance over time | 0-20 days
  calculated systemic levetiracetam clearance (based on plasma concentrations) within 48 hours of initial presentation to the neurointensive care unit and every 5 days thereafter up to 20 days

SECONDARY OUTCOMES:
Change in urinary clearance of levetiracetam and creatinine | 0-20 days
  12-hour urine collections on day 0, 5, 10, 15, and 20, calculated creatinine based on 12-hour urine collections daily for 7 days following diagnosis of vasospasm, and calculation of direct renal clearance of levetiracitam based on urine collection

CONTACTS AND LOCATIONS:
Overall Officials: Edward T Van Matre, PharmD, Principal Investigator — University of Colorado School of Pharmacy
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States